CLINICAL TRIAL: NCT04326257
Title: A Phase II Trial of Personalized Immunotherapy in Patients With Recurrent and/or Metastatic Squamous Cell Carcinoma of the Head and Neck That Have Progressed on Prior Immunotherapy
Brief Title: Personalized Immunotherapy in Patients With Recurrent /Metastatic SCCHN That Have Progressed on Prior Immunotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dan Zandberg (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Dan Zandberg, Director, Head and Neck and Thyroid Cancer Disease Sections and Co-Director, UPMC Hillman Cancer Center Head and Neck Cancer Research Program, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC 18-156
Record Dates: First submitted 2020-03-25; First posted 2020-03-30 (Actual); Results first posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: nivolumab; Relatlimab; Ipilimumab; immunotherapy; anti-PD-1; anti-PD-L1; RECIST 1.1; recurrent cancer; metastatic cancer; tumor microenvironment analysis; LAG-3; CTLA-4
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Recurrence; Neoplasm Metastasis; Diabetes Mellitus, Insulin-Dependent, 12 | interventions — Opdualag; Nivolumab; relatlimab; Ipilimumab

STUDY DESIGN:
Intervention Model Description: In this open-label, 2 parallel arms trial, RNA seq analysis via the Omniseq immune report card will be used to determine which drug (Relatlimab or Ipilimumab) will be added to Nivolumab for treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nivolumab+Relatlimab (Experimental): Nivolumab will be dosed 480mg IV q 4 weeks and Relatlimab 160mg IV q 4 weeks
  One cycle is defined as 4 weeks of treatment and both drugs are given on the same day.
  Patients will receive the prescribed therapy continuously for up to 24 cycles until progression of disease or adverse event(s) requiring treatment discontinuation.
  Interventions: Drug: Nivolumab+Relatlimab
- Nivolumab+Ipilimumab (Experimental): Nivolumab will be dosed at 3mg/kg IV q 2 weeks and Ipilimumab 1mg/kg IV q 6 weeks.
  Patients will receive four doses of Ipilimumab and the last dosage of Nivolumab 3mg/kg IV q 2 weeks will be given at the time of the 4th dose of Ipilimumab, followed 2 weeks later by Nivolumab 480 mg IV q 4 weeks. A cycle of therapy will be defined as 4 weeks of treatment. The patient will receive the prescribed therapy continuously for up to 24 cycles until progression of disease or adverse event(s) requiring treatment discontinuation.
  Interventions: Drug: Nivolumab+Ipilimumab

INTERVENTIONS:
Drug: Nivolumab+Relatlimab — IV administration of both Nivolumab and Relatlimab
  Other Names: Nivolumab: OPDIVO/ BMS-936558/ MDX1106/ ONO-4538;; Relatlimab: BMS-986016
  Arms: Nivolumab+Relatlimab
Drug: Nivolumab+Ipilimumab — IV administration of both Nivolumab and Ipilimumab
  Other Names: Nivolumab: OPDIVO/ BMS-936558/ MDX1106/ ONO-4538; Ipilimumab: YERVOY/ BMS-734016/ MDX-010
  Arms: Nivolumab+Ipilimumab

SUMMARY:
In this Phase II trial of personalized immunotherapy in R/M HNSCC, gene expression of LAG3 and CTLA4 by RNA seq will be determined to select the appropriate agent (Ipilimumab or Relatlimab) to add to Nivolumab in patients with recurrent and/or metastatic squamous cell carcinoma of the head and neck (R/M HNSCC) who have failed prior immunotherapy with anti-PD-1 or PD-L1 mAb therapy. The agent, either Ipilimumab or Relatlimab will be chosen based on the highest relevant immune gene expression (CTLA4 or LAG-3) as long as the minimum difference required is met.

DETAILED DESCRIPTION:
In this Phase II non-randomized trial, n=40 eligible patients will have tumor tissue (core or excisional/incisional) for gene expression of LAG3 and CTLA4 via RNA seq per OmniSeq Immune Report Card to determine which drug (either Relatlimab or Ipilimumab) will be added to Nivolumab for treatment. The patient will then receive the prescribed therapy continuously for up to 24 cycles (1 cycle = 28 days). The drug to be added to Nivolumab will be based on which relevant gene has the highest expression as long as the minimum difference required is met. If the minimum difference is not met than a patient will be randomized to either Nivolumab plus Relatlimab or Nivolumab plus Ipilimumab.

The patient will then receive the prescribed therapy continuously for up to 24 cycles (1 cycle = 28 days) with repeat imaging prior to every 3rd cycle until progression of disease. Response, evaluated by RECIST 1.1, with modifications to allow for continued therapy until progressive disease is confirmed if the patient is clinically stable, will be used in the trial. If the patient has confirmed progression the patient may be eligible to undergo a second biopsy and second treatment on trial. If these criteria are met the patient will then be treated with this new combination with repeat imaging prior to every 3rd cycle as per initial treatment, until progression of disease.

ELIGIBILITY:
Inclusion Criteria:

1. Recurrent and/or Metastatic squamous cell carcinoma of the head and neck that is not amenable to therapy with curative intent. Patients who refuse salvage surgery or radiation for recurrence are potentially eligible.
2. Failure of prior immunotherapy as defined as:

   1. Progression of disease on anti-PD-1 mAb or anti-PD-L1 mAb treatment in the R/M setting.
   2. Both patients that have received platinum based chemotherapy prior or have not yet received platinum based chemotherapy are eligible.
3. Patients cannot have received more than 3 total lines of prior systemic therapy in the recurrent/metastatic setting.
4. ECOG performance status of 0-1
5. Have at least one measurable area of disease (Target Lesion) based on RECIST 1.1.
6. Provide adequate tissue (core or incisional/excisional biopsy) prior to starting study for analysis for gene expression of LAG3 and CTLA4 per OmniSeq Immune Report Card. FNA is not adequate. Archival tissue can only be used if it was obtained in the recurrent/metastatic setting and there has been no subsequent cancer treatment after that tissue was obtained.
7. Life expectancy of at least 12 weeks based on investigator estimate.
8. Age ≥ 18 years old
9. LVEF assessment with documented LVEF ≥50% by either TTE or MUGA (TTE preferred test) within 6 months from first study drug administration
10. Patients must have normal organ and marrow function as defined below:

    * absolute neutrophil count ≥1,500/mcL
    * platelets ≥100,000/mcL
    * total bilirubin ≤ institutional upper limit of normal (ULN)
    * AST(SGOT)/ALT(SGPT) ≤2.5 x institutional ULN
    * creatinine ≤ institutional ULN

    OR

    - glomerular filtration rate ≥40 mL/min/1.73 m2 for patients with creatinine levels. (GFR) above institutional normal.
11. Female subjects of childbearing potential should have a negative urine or serum pregnancy within 1 days prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
12. Female subjects of childbearing potential should be willing to use 1 methods of birth control or abstain from heterosexual activity for the course of the study through 5 months after the last dose of study medication. Women of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
13. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 7 months after the last dose of study therapy.
14. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. SCC of salivary gland origin or cutaneous SCC of the head and neck. HNSCC of unknown origin ARE eligible.
2. Patients who received Ipilimumab or Relatlimab in the recurrent/metastatic setting will be excluded.
3. Is currently participating in or has participated in a study of an investigational agent or used an investigational device within 2 weeks of the first dose of treatment.
4. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (equivalent of >10 mg of prednisone) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
5. Has had a prior monoclonal antibody, chemotherapy, or targeted small molecule therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier (alopecia is an exception). Note: Subjects with ≤ Grade 2 neuropathy, ototoxicity, hypothyroidism or hyperthyroidism, are an exception to this criterion and qualify for the study.
6. History of other malignancy within 3 years with the exception of prior HNSCC, adequately treated basal cell or squamous cell skin cancer, or carcinoma of the cervix.
7. Has an active autoimmune disease requiring systemic immunosuppressive treatment within the past 3 months. Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic therapy or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study.
8. Uncontrolled or significant cardiovascular disease including, but not limited to, any of the following:

   1. Myocardial infarction (MI) or stroke/transient ischemic attack (TIA) within the 6 months prior to consent;
   2. Uncontrolled angina within the 3 months prior to consent;
   3. Any history of clinically significant arrhythmias (such as ventricular tachycardia, ventricular fibrillation, torsades de pointes, or poorly controlled atrial fibrillation);
   4. QTc prolongation > 480 msec;
   5. History of other clinically significant cardiovascular disease (i.e., cardiomyopathy, congestive heart failure with New York Heart Association [NYHA] functional classification III-IV, pericarditis, significant pericardial effusion, significant coronary stent occlusion, poorly controlled deep venous thrombosis, etc.);
   6. Cardiovascular disease-related requirement for daily supplemental oxygen
   7. History of two or more MIs OR two or more coronary revascularization procedures
   8. Subjects with history of myocarditis, regardless of etiology.
9. A confirmed history of encephalitis, meningitis, or uncontrolled seizures in the year prior to informed consent
10. Subjects with history of life-threatening toxicity related to prior immune therapy (eg. anti-CTLA-4 or anti-PD-1/PD-L1 treatment or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways) except those that are unlikely to re-occur with standard countermeasures (eg, hormone replacement after endocrinopathy).
11. Troponin T (TnT) or I (TnI) > 2 × institutional ULN. Subjects with TnT or TnI levels between > 1 to 2 × ULN will be permitted if repeat levels within 24 hours are ≤1 x ULN. If TnT or TnI levels are >1 to 2 × ULN within 24 hours, the subject may undergo a cardiac evaluation and be considered for treatment based on the discretion of the PI. When repeat levels within 24 hours are not available, a repeat test should be conducted as soon as possible. If TnT or TnI repeat levels beyond 24 hours are < 2 x ULN, the subject may undergo a cardiac evaluation and be considered for treatment, based on the discretion of the PI.
12. Has a history of non-infectious pneumonitis that required steroids, evidence of interstitial lung disease, or currently active non-infectious pneumonitis.
13. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
14. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
15. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 24 weeks after the last dose of trial treatment.
16. Has a history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
17. Has active Hepatitis B or Hepatitis C
18. Has a history of a solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-05-14 (Actual); Primary Completion 2023-08-12 (Actual); Study Completion 2024-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan P Zandberg, MD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Selected Treatment; Randomized Treatment: Nivolumab+Relatlimab:
  Nivolumab will be dosed 480mg IV q 4 weeks and Relatlimab 160mg IV q 4 weeks One cycle is defined as 4 weeks of treatment and both drugs are given on the same day.
  Patients will receive the prescribed therapy continuously for up to 24 cycles until progression of disease or adverse event(s) requiring treatment discontinuation.
  Or,
  Nivolumab+Ipilimumab: IV administration of both Nivolumab and Ipilimumab Nivolumab will be dosed at 3mg/kg IV q 2 weeks and Ipilimumab 1mg/kg IV q 6 weeks.
  Patients will receive four doses of Ipilimumab and the last dosage of Nivolumab 3mg/kg IV q 2 weeks will be given at the time of the 4th dose of Ipilimumab, followed 2 weeks later by Nivolumab 480 mg IV q 4 weeks. A cycle of therapy will be defined as 4 weeks of treatment. The patient will receive the prescribed therapy continuously for up to 24 cycles until progression of disease or adverse event(s) requiring treatment discontinuation.
Period: Overall Study
Arm/Group | Selected Treatment | Randomized Treatment
Started | 7 | 13
Nivolumab+Relatlimab | 7 | 6
Nivolumab+Ipilimumab | 0 | 7
Completed | 7 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: It was pre-specified to report data per the two groups of interest, "selected" or "randomized," without specific drug combinations.
Groups:
- Selected Treatment; Randomized Treatment: Nivolumab+Relatlimab: IV administration of both Nivolumab and Relatlimab Nivolumab will be dosed 480mg IV q 4 weeks and Relatlimab 160mg IV q 4 weeks One cycle is defined as 4 weeks of treatment and both drugs are given on the same day.
  Patients will receive the prescribed therapy continuously for up to 24 cycles until progression of disease or adverse event(s) requiring treatment discontinuation.
  Or,
  Nivolumab+Ipilimumab: IV administration of both Nivolumab and Ipilimumab Nivolumab will be dosed at 3mg/kg IV q 2 weeks and Ipilimumab 1mg/kg IV q 6 weeks.
  Patients will receive four doses of Ipilimumab and the last dosage of Nivolumab 3mg/kg IV q 2 weeks will be given at the time of the 4th dose of Ipilimumab, followed 2 weeks later by Nivolumab 480 mg IV q 4 weeks. A cycle of therapy will be defined as 4 weeks of treatment. The patient will receive the prescribed therapy continuously for up to 24 cycles until progression of disease or adverse event(s) requiring treatment discontinuation.
- Total: Total of all reporting groups
Arm/Group | Selected Treatment | Randomized Treatment | Total
Number analyzed (Participants) | 7 | 13 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.86 (9.974) | 63.62 (7.633) | 63.35 (8.267)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 7 | 11 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 13 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 13 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Probability of Objective Response (OR) - Selected Treatment
Description: The probability of response to therapy in patients who have progressed on prior immunotherapy. Per Response Evaluation Criteria in Solid Tumors (RECIST v1.1) Complete Response (CR) is disappearance of all target and non-target lesions; Partial Response (PR) is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From start of treatment, up to 36 months
Population: Treated patients who were radiologically evaluable. It was pre-specified to report data per the two groups of interest, "selected" or "randomized," without specific drug combinations.
Measure: Number; unit: percentage of patients
Arm/Group | Selected Treatment
Number analyzed (Participants) | 7
percentage of patients | 0

2. Secondary Outcome: Probability of Objective Response (OR) - Randomized Treatment
Description: as for outcome 1
Time Frame: From start of treatment, up to 36 months
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | Randomized Treatment
Number analyzed (Participants) | 7
percentage of patients | 0

3. Secondary Outcome: Disease Control Rate (DCR)
Description: The percent probability of not experiencing disease progression in patients regardless of selected/randomized treatment. Per Response Evaluation Criteria in Solid Tumors (RECIST v1.1) Complete Response (CR) is disappearance of all target and non-target lesions; Partial Response (PR) is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters; Stable Disease (SD) is neither sufficient decrease (target lesions) to qualify as a PR or sufficient increase to qualify as PD. Incomplete Response/Stable Disease (SD) is the persistence of one or more non-target lesions.
Time Frame: From start of treatment, up to 36 months
Population: Treated patients evaluable for radiologic response. It was pre-specified to report data per the two groups of interest, "selected" or "randomized," without specific drug combinations.
Measure: Number (95% Confidence Interval); unit: percent probability of participants
Arm/Group | Selected Treatment | Randomized Treatment
Number analyzed (Participants) | 6 | 12
percent probability of participants | 33.3 [9.7 to 70.0] | 25.0 [8.9 to 53.2]

4. Secondary Outcome: Progression-free Survival (PFS)
Description: The length of time from the start of treatment that patients live with disease that does not progress per Response Evaluation Criteria in Solid Tumors (RECIST v1.1) in patients who have progressed on prior immunotherapy. Per RECIST, Progressive Disease (PD) is defined as at least a 20% increase in the sum of the diameters of target lesions compared to baseline sum of target lesions, or any new lesions.It also includes the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: From start of treatment up to 36 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Selected Treatment; Randomized Treatment: Nivolumab+Relatlimab: IV administration of both Nivolumab and Relatlimab Nivolumab will be dosed 480mg IV q 4 weeks and Relatlimab 160mg IV q 4 weeks One cycle is defined as 4 weeks of treatment and both drugs are given on the same day.
  Patients will receive the prescribed therapy continuously for up to 24 cycles until progression of disease or adverse event(s) requiring treatment discontinuation.
  Nivolumab+Ipilimumab: IV administration of both Nivolumab and Ipilimumab Nivolumab will be dosed at 3mg/kg IV q 2 weeks and Ipilimumab 1mg/kg IV q 6 weeks.
  Patients will receive four doses of Ipilimumab and the last dosage of Nivolumab 3mg/kg IV q 2 weeks will be given at the time of the 4th dose of Ipilimumab, followed 2 weeks later by Nivolumab 480 mg IV q 4 weeks. A cycle of therapy will be defined as 4 weeks of treatment. The patient will receive the prescribed therapy continuously for up to 24 cycles until progression of disease or adverse event(s) requiring treatment discontinuation.
Arm/Group | Selected Treatment | Randomized Treatment
Number analyzed (Participants) | 6 | 11
Days | 52.00 [31.60 to 72.40] | 53.00 [50.92 to 55.09]

5. Secondary Outcome: Overall Survival (OS)
Description: The length of time from the start of treatment that patients remain alive, in patients who have progressed on prior immunotherapy.
Time Frame: From start of treatment, up to 36 months
Population: All enrolled patients. It was pre-specified to report data per the two groups of interest, "selected" or "randomized," without specific drug combinations.
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Randomized Treatment: Nivolumab will be dosed at 3mg/kg IV q 2 weeks and Ipilimumab 1mg/kg IV q 6 weeks.
  Patients will receive four doses of Ipilimumab and the last dosage of Nivolumab 3mg/kg IV q 2 weeks will be given at the time of the 4th dose of Ipilimumab, followed 2 weeks later by Nivolumab 480 mg IV q 4 weeks. A cycle of therapy will be defined as 4 weeks of treatment. The patient will receive the prescribed therapy continuously for up to 24 cycles until progression of disease or adverse event(s) requiring treatment discontinuation.
  Nivolumab+Ipilimumab: IV administration of both Nivolumab and Ipilimumab
Arm/Group | Selected Treatment | Randomized Treatment
Number analyzed (Participants) | 5 | 6
Days | 166.00 [22.92 to 309.08] | 164.00 [0.00 to 379.60]

6. Secondary Outcome: Duration of Disease Control
Description: Mean number of months that patients who had Stable Disease experienced disease control. Per Response Evaluation Criteria in Solid Tumors (RECIST v1.1) Stable Disease (SD) is neither sufficient decrease (target lesions) to qualify as a PR or sufficient increase to qualify as PD. Incomplete Response/Stable Disease (SD) is the persistence of one or more non-target lesions.
Time Frame: From start of treatment, up to 36 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Selected Treatment | Randomized Treatment
Number analyzed (Participants) | 2 | 3
Days | 133.50 (122.33) | 97.67 (81.82)

7. Secondary Outcome: Adverse Events Per Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Description: Adverse Events possibly, probably or definitely related to study treatment per Common Terminology Criteria for Adverse Events (CTCAE) v5.0 experienced.
Time Frame: From start of treatment, up to 36 months
Population: Distinct number of treated patients. It was pre-specified to report data per the two groups of interest, "selected" or "randomized," without specific drug combinations.
Measure: Number; unit: patients
Groups:
- Nivolumab+Relatlimab: Nivolumab will be dosed 480mg IV q 4 weeks and Relatlimab 160mg IV q 4 weeks
  One cycle is defined as 4 weeks of treatment and both drugs are given on the same day.
  Patients will receive the prescribed therapy continuously for up to 24 cycles until progression of disease or adverse event(s) requiring treatment discontinuation.
  Nivolumab+Relatlimab: IV administration of both Nivolumab and Relatlimab
- Nivolumab+Ipilimumab: Nivolumab will be dosed at 3mg/kg IV q 2 weeks and Ipilimumab 1mg/kg IV q 6 weeks.
  Patients will receive four doses of Ipilimumab and the last dosage of Nivolumab 3mg/kg IV q 2 weeks will be given at the time of the 4th dose of Ipilimumab, followed 2 weeks later by Nivolumab 480 mg IV q 4 weeks. A cycle of therapy will be defined as 4 weeks of treatment. The patient will receive the prescribed therapy continuously for up to 24 cycles until progression of disease or adverse event(s) requiring treatment discontinuation.
  Nivolumab+Ipilimumab: IV administration of both Nivolumab and Ipilimumab
Arm/Group | Nivolumab+Relatlimab | Nivolumab+Ipilimumab
Number analyzed (Participants) | 13 | 7
patients
  Alanine aminotransferase increased | 3 | 1
  Alkaline phosphatase increased | 2 | 0
  Anemia | 2 | 2
  Anorexia | 1 | 0
  Aspartate aminotransferase increased | 3 | 1
  PACs on EKG | 1 | 0
  Cough | 0 | 1
  Creatinine increased | 1 | 0
  Fatigue | 2 | 1
  Hyperglycemia | 1 | 0
  Hypoalbuminemia | 1 | 0
  Hyponatremia | 2 | 1
  Hypophosphatemia | 2 | 0
  Lymphocyte count decreased | 3 | 1
  Platelet count decreased | 1 | 1
  psoriasis | 1 | 0
  Tumor hemorrhage | 1 | 0
  Vomiting | 1 | 1
  Weight loss | 0 | 1
  Rash maculo-papular | 0 | 1
  Pneumonitis | 0 | 1
  Diarrhea | 0 | 2
  Flushing | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse Events data were collected for up to 36 months. All-Cause Mortality data was collected for up to 46 months.
Description: It was pre-specified to report data per the two groups of interest, "selected" or "randomized," without specific drug combinations.
Groups:
- Nivolumab+Relatlimab: Nivolumab will be dosed 480mg IV q 4 weeks and Relatlimab 160mg IV q 4 weeks
  One cycle is defined as 4 weeks of treatment and both drugs are given on the same day.
  Patients received the prescribed therapy continuously for up to 24 cycles until progression of disease or adverse event(s) requiring treatment discontinuation.
  Nivolumab+Relatlimab: IV administration of both Nivolumab and Relatlimab
- Nivolumab+Ipilimumab: Nivolumab will be dosed at 3mg/kg IV q 2 weeks and Ipilimumab 1mg/kg IV q 6 weeks.
  Patients received four doses of Ipilimumab and the last dosage of Nivolumab 3mg/kg IV q 2 weeks will be given at the time of the 4th dose of Ipilimumab, followed 2 weeks later by Nivolumab 480 mg IV q 4 weeks.
  One cycle of therapy will be defined as 4 weeks of treatment.
  Patients received the prescribed therapy continuously for up to 24 cycles until progression of disease or adverse event(s) requiring treatment discontinuation.
  Nivolumab+Ipilimumab: IV administration of both Nivolumab and Ipilimumab
Arm/Group | Nivolumab+Relatlimab | Nivolumab+Ipilimumab
All-Cause Mortality (participants affected / at risk) | 12/13 | 4/7
Serious Adverse Events (participants affected / at risk) | 11/13 | 6/7
Other Adverse Events (participants affected / at risk) | 10/13 | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab+Relatlimab (N=13) | Nivolumab+Ipilimumab (N=7)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 1
Agitation (Psychiatric disorders) | 0 | 0
Alanine aminotransferase increased (Investigations) | 4 | 1
Alkaline phosphatase increased (Investigations) | 3 | 2
Anemia (Blood and lymphatic system disorders) | 10 | 6
Anorexia (Metabolism and nutrition disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
Bone marrow hypocellular (Blood and lymphatic system disorders) | 1 | 0
Cardiac disorders - Other, specifyCoronary artery disease (Cardiac disorders) | 1 | 0
Cardiac disorders - Other, specifyPACs on EKG (Cardiac disorders) | 1 | 0
Cardiac disorders - Other, specifyright bundle branch block (Cardiac disorders) | 1 | 0
Cardiac troponin I increased (Investigations) | 1 | 0
Cholesterol high (Investigations) | 1 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Confusion (Psychiatric disorders) | 0 | 0
Constipation (Gastrointestinal disorders) | 4 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Creatinine increased (Investigations) | 3 | 1
Depression (Psychiatric disorders) | 1 | 3
Diarrhea (Gastrointestinal disorders) | 3 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 3
Dysarthria (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Ear and labyrinth disorders - Other, specifyR ear drainage ottorrhea (Ear and labyrinth disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 0
Facial pain (General disorders) | 2 | 0
Fatigue (General disorders) | 6 | 4
Fever (General disorders) | 1 | 0
Gait disturbance (General disorders) | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 | 2
Gastrointestinal disorders - Other, specifyDiverticulitis (Gastrointestinal disorders) | 0 | 0
Gastrointestinal disorders - Other, specifyDuodenitis (Gastrointestinal disorders) | 1 | 0
General disorders and administration site conditions - Other, specifyFailure to thrive (General disorders) | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 1
Hearing impaired (Ear and labyrinth disorders) | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 5 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hyperlipidemia (Metabolism and nutrition disorders) | 1 | 1
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0
Hypertension (Vascular disorders) | 4 | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 4 | 1
Hyponatremia (Metabolism and nutrition disorders) | 6 | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 4 | 0
Hypotension (Vascular disorders) | 1 | 1
Hypothyroidism (Endocrine disorders) | 4 | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Immune system disorders - Other, specifyCeliacs disease (Immune system disorders) | 1 | 0
Infections and infestations - Other, specifyRight neck (Infections and infestations) | 1 | 0
Infections and infestations - Other, specifyThrush (Infections and infestations) | 1 | 1
Injury, poisoning and procedural complications - Other, specifyLeft neck wound, biopsy site (Injury, poisoning and procedural complications) | 1 | 0
Injury, poisoning and procedural complications - Other, specifyRadiation fibrosis (Injury, poisoning and procedural complications) | 1 | 0
INR increased (Investigations) | 2 | 0
Insomnia (Psychiatric disorders) | 2 | 2
Investigations - Other, specifyalbumin decrease (Investigations) | 1 | 0
Investigations - Other, specifyBlood bicarbonate decrease (Investigations) | 1 | 0
Investigations - Other, specifyIncreased LDH (Investigations) | 1 | 0
Investigations - Other, specifyVitamin D deficiency (Investigations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Lymphedema (Vascular disorders) | 1 | 0
Lymphocyte count decreased (Investigations) | 5 | 3
Metabolism and nutrition disorders - Other, specifyHyperphosphatemia (Metabolism and nutrition disorders) | 1 | 0
Metabolism and nutrition disorders - Other, specifyType II Diabetes (Metabolism and nutrition disorders) | 2 | 0
Musculoskeletal and connective tissue disorder - Other, specifymuscle cramp (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specifyosteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specifyosteomyelitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specifyBone Metastases (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specifyLipomas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Nervous system disorders - Other, specifydestruction of facial nerves (Nervous system disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 1
Oral pain (Gastrointestinal disorders) | 3 | 2
Pain (General disorders) | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 1
Platelet count decreased (Investigations) | 3 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, specifyCOPD (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory, thoracic and mediastinal disorders - Other, specifyParalyzed diaphragm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, specifyPneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, specifytrach secretions (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sepsis (Infections and infestations) | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 2
Sinus tachycardia (Cardiac disorders) | 2 | 0
Skin and subcutaneous tissue disorders - Other, specifypharyngeal erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Skin and subcutaneous tissue disorders - Other, specifypsoriasis (Skin and subcutaneous tissue disorders) | 0 | 0
Skin and subcutaneous tissue disorders - Other, specifySeborrhea capitis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Stomach pain (Gastrointestinal disorders) | 1 | 0
Surgical and medical procedures - Other, specifyL sided neck dissection (Surgical and medical procedures) | 0 | 0
Surgical and medical procedures - Other, specifyThymectomy of mediastinal Mass (Surgical and medical procedures) | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 2 | 0
Tremor (Nervous system disorders) | 1 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Vascular disorders - Other, specifyDeep vein thrombosis (Vascular disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Weight loss (Investigations) | 2 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
White blood cell decreased (Investigations) | 3 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab+Relatlimab (N=13) | Nivolumab+Ipilimumab (N=7)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 1
Agitation (Psychiatric disorders) | 0 | 0
Alanine aminotransferase increased (Investigations) | 4 | 1
Alkaline phosphatase increased (Investigations) | 3 | 2
Anemia (Blood and lymphatic system disorders) | 10 | 6
Anorexia (Metabolism and nutrition disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
Bone marrow hypocellular (Blood and lymphatic system disorders) | 1 | 0
Cardiac disorders - Other, specifyCoronary artery disease (Cardiac disorders) | 1 | 0
Cardiac disorders - Other, specifyPACs on EKG (Cardiac disorders) | 1 | 0
Cardiac disorders - Other, specifyright bundle branch block (Cardiac disorders) | 1 | 0
Cardiac troponin I increased (Investigations) | 1 | 0
Cholesterol high (Investigations) | 1 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Confusion (Psychiatric disorders) | 0 | 0
Constipation (Gastrointestinal disorders) | 4 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Creatinine increased (Investigations) | 3 | 1
Depression (Psychiatric disorders) | 1 | 3
Diarrhea (Gastrointestinal disorders) | 3 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 3
Dysarthria (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Ear and labyrinth disorders - Other, specifyR ear drainage ottorrhea (Ear and labyrinth disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 0
Facial pain (General disorders) | 2 | 0
Fatigue (General disorders) | 6 | 4
Fever (General disorders) | 1 | 0
Gait disturbance (General disorders) | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 | 2
Gastrointestinal disorders - Other, specifyDiverticulitis (Gastrointestinal disorders) | 0 | 0
Gastrointestinal disorders - Other, specifyDuodenitis (Gastrointestinal disorders) | 1 | 0
General disorders and administration site conditions - Other, specifyFailure to thrive (General disorders) | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 1
Hearing impaired (Ear and labyrinth disorders) | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 5 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hyperlipidemia (Metabolism and nutrition disorders) | 1 | 1
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0
Hypertension (Vascular disorders) | 4 | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 4 | 1
Hyponatremia (Metabolism and nutrition disorders) | 6 | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 4 | 0
Hypotension (Vascular disorders) | 1 | 1
Hypothyroidism (Endocrine disorders) | 4 | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Immune system disorders - Other, specifyCeliacs disease (Immune system disorders) | 1 | 0
Infections and infestations - Other, specifyRight neck (Infections and infestations) | 1 | 0
Infections and infestations - Other, specifyThrush (Infections and infestations) | 1 | 1
Injury, poisoning and procedural complications - Other, specifyLeft neck wound, biopsy site (Injury, poisoning and procedural complications) | 1 | 0
Injury, poisoning and procedural complications - Other, specifyRadiation fibrosis (Injury, poisoning and procedural complications) | 1 | 0
INR increased (Investigations) | 2 | 0
Insomnia (Psychiatric disorders) | 2 | 2
Investigations - Other, specifyalbumin decrease (Investigations) | 1 | 0
Investigations - Other, specifyBlood bicarbonate decrease (Investigations) | 1 | 0
Investigations - Other, specifyIncreased LDH (Investigations) | 1 | 0
Investigations - Other, specifyVitamin D deficiency (Investigations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Lymphedema (Vascular disorders) | 1 | 0
Lymphocyte count decreased (Investigations) | 5 | 3
Metabolism and nutrition disorders - Other, specifyHyperphosphatemia (Metabolism and nutrition disorders) | 1 | 0
Metabolism and nutrition disorders - Other, specifyType II Diabetes (Metabolism and nutrition disorders) | 2 | 0
Musculoskeletal and connective tissue disorder - Other, specifymuscle cramp (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specifyosteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specifyosteomyelitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specifyBone Metastases (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specifyLipomas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Nervous system disorders - Other, specifydestruction of facial nerves (Nervous system disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 1
Oral pain (Gastrointestinal disorders) | 3 | 2
Pain (General disorders) | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 1
Platelet count decreased (Investigations) | 3 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, specifyCOPD (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory, thoracic and mediastinal disorders - Other, specifyParalyzed diaphragm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, specifyPneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, specifytrach secretions (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sepsis (Infections and infestations) | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 2
Sinus tachycardia (Cardiac disorders) | 2 | 0
Skin and subcutaneous tissue disorders - Other, specifypharyngeal erythema (Skin and subcutaneous tissue disorders) | 1 | 0
psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin and subcutaneous tissue disorders - Other, specifySeborrhea capitis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Stomach pain (Gastrointestinal disorders) | 1 | 0
Surgical and medical procedures - Other, specifyL sided neck dissection (Surgical and medical procedures) | 0 | 0
Surgical and medical procedures - Other, specifyThymectomy of mediastinal Mass (Surgical and medical procedures) | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 2 | 0
Tremor (Nervous system disorders) | 1 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Vascular disorders - Other, specifyDeep vein thrombosis (Vascular disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Weight loss (Investigations) | 2 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
White blood cell decreased (Investigations) | 3 | 1
PACs on EKG (Cardiac disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Flushing (Vascular disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-04): https://cdn.clinicaltrials.gov/large-docs/57/NCT04326257/Prot_SAP_000.pdf